CLINICAL TRIAL: NCT00009919
Title: Phase II Study of SU5416 (NSC 696819) for Patients With Progressive Metastatic Renal Cancer Failing Prior Biologic Therapy or 5-Fluorouracil Containing Regimens
Brief Title: SU5416 in Treating Patients With Metastatic Kidney Cancer That Has Not Responded to Previous Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02373; ID99-291; N01CM17003 (NIH); CDR0000068424 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-02-02; First posted 2004-01-01 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Semaxinib

ARMS (1):
- Treatment (semaxanib) (Experimental): Patients receive SU5416 IV over 1 hour twice weekly. Treatment continues every 6 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with CR receive an additional 6 months of therapy after achieving CR.
  Interventions: Drug: semaxanib

INTERVENTIONS:
Drug: semaxanib — Given IV
  Other Names: semoxind; SU5416; Sugen 5416

SUMMARY:
Phase II trial to study the effectiveness of SU5416 in treating patients who have metastatic kidney cancer that has not responded to previous therapy with interleukin-2. SU5416 may stop the growth of kidney cancer by stopping blood flow to the tumor

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the clinical activity of SU5416 in patients with progressive metastatic renal cancer failing prior biologic therapy or fluorouracil-containing regimens.

II. Determine the changes in tumor perfusion in patients treated with this regimen.

III. Determine the time to progression and survival in patients treated with this regimen.

OUTLINE:

Patients receive SU5416 IV over 1 hour twice weekly. Treatment continues every 6 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with complete response (CR) receive an additional 6 months of therapy after achieving CR.

Patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic renal cell carcinoma
* Prior removal of primary tumors
* Bidimensionally measurable disease

  * Bone-only disease is not considered measurable
* Progressive disease following no more than 2 prior biologic therapy (e.g.,interleukin-2, interferon alfa, vaccine, or dendritic cell therapy) orfluorouracil-containing (single-agent or in combination therapy) regimens
* No known history of CNS metastasis unless all of the following are true:

  * Previously treated
  * Neurologically stable
  * No requirement for IV steroids or anticonvulsants
  * No requirement for oral steroids and no evidence of active or residual CNS disease on CT scan or MRI
* Negative brain scan (CT scan or MRI) required if neurologic signs or symptoms suggestive of CNS metastasis present
* Performance status - Zubrod 0-2
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* SGPT no greater than 2.5 times upper limit of normal
* PT and PTT normal
* Fibrinogen normal
* D-Dimer assay normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* See Surgery
* No active congestive heart failure
* No uncontrolled angina
* No myocardial infarction or severe/unstable angina within the past 6 months
* No uncontrolled hypertension
* No uncompensated coronary artery disease on electrocardiogram or physical examination
* No severe peripheral vascular disease
* No deep vein or arterial thrombosis within the past 3 months
* No pulmonary embolism within the past 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent serious infection
* No overt psychosis, mental disability, or incompetence
* No diabetes mellitus
* No other prior malignancy within the past 5 years except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No hypersensitivity or allergic reaction to paclitaxel
* See Disease Characteristics
* No other concurrent anti-cancer biologic therapy
* See Disease Characteristics
* No concurrent anti-cancer chemotherapy
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No sole indicator lesion within the previously irradiated port
* No concurrent anti-cancer radiotherapy
* See Disease Characteristics
* At least 4 weeks since prior major surgery and recovered
* At least 1 year since prior bypass surgery for atherosclerotic coronary artery disease
* No concurrent surgery for cancer
* No other investigational drugs (e.g., analgesics or antiemetics) for at least 28 days prior to and after study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2000-12; Primary Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Rate of progression-free events | 6 months
  Estimated with associated confidence intervals using standard methods such as chi-square and Fisher's exact tests.
Objective response rate | Up to 3 years
  Estimated with associated confidence intervals using standard methods such as chi-square and Fisher's exact tests.

SECONDARY OUTCOMES:
Survival | Up to 3 years
  Analyzed using Kaplan Meier curves and Cox proportional hazards models.
Time to disease progression | Up to 3 years
  Analyzed using Kaplan Meier curves and Cox proportional hazards.
Time to treatment failure | Up to 3 years
  Analyzed using Kaplan Meier curves and Cox proportional hazards.
Duration of response | Up to 3 years
  Analyzed using Kaplan Meier curves and Cox proportional hazards.

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Siefker-Radtke, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States